CLINICAL TRIAL: NCT03182504
Title: A Non-Randomized, Open Label, One Treatment, One Group Study to Investigate the Intrapulmonary Lung Penetration of RO7079901 in Healthy Volunteers
Brief Title: A Study to Investigate the Intrapulmonary Lung Penetration of Nacubactam in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP39750; 2016-004478-16 (EudraCT Number)
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Gram-negative Bacterial Infections
MeSH Terms: conditions — Gram-Negative Bacterial Infections | interventions — nacubactam; Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nacubactam Plus Meropenem (Experimental): Participants will receive a single dose of nacubactam co-administered with meropenem.
  Interventions: Drug: nacubactam; Drug: meropenem

INTERVENTIONS:
Drug: nacubactam — Participants will receive a single 2000 milligram (mg) intravenous (IV) infusion of nacubactam over 1.5 hours.
  Other Names: RO7079901
Drug: meropenem — Participants will receive a single 2000 mg IV infusion of meropenem over 1.5 hours.
  Other Names: Merrem

SUMMARY:
The purpose of this study is to characterize the intrapulmonary penetration of nacubactam in healthy volunteers. Nacubactam is a novel non-beta-lactam beta-lactamase inhibitor being developed as a combination therapy with the beta-lactam meropenem for the treatment of serious gram-negative bacterial infections. Adult male and female healthy participants will receive a single intravenous infusion of nacubactam co-administered with meropenem and then undergo a bronchoalveolar lavage (BAL) procedure to collect lung epithelial lining fluid (ELF) for measurement of intrapulmonary concentrations of nacubactam and meropenem.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years of age, inclusive
* Healthy, as judged by the Investigator and defined by the absence of evidence of any active or clinically significant chronic disease identified from a detailed medical and surgical history, physical examination including vital signs and 12-lead electrocardiogram (ECG), and laboratory safety test results
* Body mass index (BMI) within the range 18-30 kilogram per square meter (kg/m^2),inclusive
* Non-smoker, or former smoker who has abstained from smoking for at least 6 months
* Negative pregnancy test and agreement to comply with measures to prevent pregnancy in women
* Refrain from sperm donation and agreement to comply with measures to prevent pregnancy in partner of childbearing potential for men

Exclusion Criteria:

* History of asthma or clinically significant lung disease
* Any condition which contraindicates a BAL procedure
* History of clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardiovascular, endocrinological, hematological, dermatological, immunological or allergic disease, metabolic disorder, cancer or cirrhosis
* Clinically significant change in health status, as judged by the Investigator, or any major illness within the four weeks before screening, or clinically significant acute infection or febrile illness within the 14 days before screening
* History of epilepsy (or known seizure disorder), brain lesions or other significant neurological disorders
* Participation in any other clinical study involving an investigational medicinal product or device within 3 months before screening
* Known history of clinically significant hypersensitivity or urticaria, or severe allergic reaction to any drug, in particular antibiotics
* Donation or loss of over 500 milliliter (mL) of blood within the three months before screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
Epithelial Lining Fluid (ELF) Concentration of Nacubactam to Plasma Concentration of Nacubactam Ratio | At 2, 3, 4, 6 and 8 hours after study drug administration
  The ELF to plasma ratio will be calculated from the concentration of nacubactam in ELF and plasma as a measure of the intrapulmonary penetration of nacubactam in healthy participants.

SECONDARY OUTCOMES:
ELF Concentration of Meropenem to Plasma Concentration of Meropenem Ratio | At 2, 3, 4, 6 and 8 hours after study drug administration
  The ELF to plasma ratio will be calculated from the concentration of meropenem in ELF and plasma as a measure of the intrapulmonary penetration of meropenem in healthy participants..
Area Under the Plasma Concentration-Time Curve from time 0 to 8 hours (AUC0-8) of Nacubactam in ELF | At 2, 3, 4, 6 and 8 hours after study drug administration
Maximum Concentration (Cmax) of Nacubactam in ELF | At 2, 3, 4, 6 and 8 hours after study drug administration
Area Under the Plasma Concentration-Time Curve from Time 0 to 8 Hours (AUC0-8) of Nacubactam in Blood Plasma | At 0, 0.75, 1.5, 2, 3, 4, 6 and 8 hours after study drug administration
Maximum Concentration (Cmax) of Nacubactam in Blood Plasma | At 0, 0.75, 1.5, 2, 3, 4, 6 and 8 hours after study drug administration
Time to Reach the Maximum Plasma Concentration (Tmax) of Nacubactam | At 0, 0.75, 1.5, 2, 3, 4, 6 and 8 hours after study drug administration
Clearance (CL) of Nacubactam | At 0, 0.75, 1.5, 2, 3, 4, 6 and 8 hours after study drug administration
Volume of Distribution of the Central Compartment (Vc) of Nacubactam | At 0, 0.75, 1.5, 2, 3, 4, 6 and 8 hours after study drug administration
Volume of Distribution at Steady-State (Vss) of Nacubactam | At 0, 0.75, 1.5, 2, 3, 4, 6 and 8 hours after study drug administration
Area Under the Plasma Concentration-Time Curve from Time 0 to 8 Hours (AUC0-8) of Meropenem in ELF | At 2, 3, 4, 6 and 8 hours after study drug administration
Maximum Concentration (Cmax) of Meropenem in ELF | At 2, 3, 4, 6 and 8 hours after study drug administration
Area Under the Plasma Concentration-Time Curve from Time 0 to 8 hours (AUC0-8) of Meropenem in Blood Plasma | At 0, 0.75, 1.5, 2, 3, 4, 6 and 8 hours after study drug administration
Maximum Concentration (Cmax) of Meropenem in Blood Plasma | At 0, 0.75, 1.5, 2, 3, 4, 6 and 8 hours after study drug administration
Time to Reach the Maximum Plasma Concentration (Tmax) of Meropenem | At 0, 0.75, 1.5, 2, 3, 4, 6 and 8 hours after study drug administration
Clearance (CL) of Meropenem | At 0, 0.75, 1.5, 2, 3, 4, 6 and 8 hours after study drug administration
Volume of Distribution of the Central Compartment (Vc) of Meropenem | At 0, 0.75, 1.5, 2, 3, 4, 6 and 8 hours after study drug administration
Volume of Distribution at Steady-State (Vss) of Meropenem | At 0, 0.75, 1.5, 2, 3, 4, 6 and 8 hours after study drug administration
Number of Participants with Adverse Events | From baseline up to 14 days after study drug administration
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Pulmonary Associates Clinical Trials (PACT), Phoenix, Arizona, United States